CLINICAL TRIAL: NCT00538226
Title: To Evaluate the Increase of Local Circulation in the Leg Using the Flowaid Device
Brief Title: Evaluation of the Effect of the Flowaid Device in Increasing Local Circulation in the Leg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rosenblum, Jonathan I., DPM (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: tali725
Record Dates: First submitted 2007-09-29; First posted 2007-10-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2008-03

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: External Electric Muscle Stimulation

SUMMARY:
This is an open label pilot study to evaluate the efficacy and the safety of the Flowaid device in increasing local circulation in the legs.

15 patients with a diagnosis of Peripheral Vascular Disease will be enrolled in this study. They will recieve tratment with the Flowaid device and monitored continuously by means of Laser Doppler Flowmetry as well as by tcPO2 and Digital Thermography. Subjective data will also be collected.

DETAILED DESCRIPTION:
This is a 15 patient pilot study to evaluate efficacy and safety of use of the Flowaid device in increasing local circulation in the legs of patients with Peripheral Vascular Disease. Patients will be evaluated and scored prior to treatment and then treated with the Flowaid device for a period of two hours. During the treatment period patients will be continuously monitored by digital thermograph as well as by tcPO2 and Laser Doppler Flowmetry. Patients will also be monitored for a brief period immediately after cessation of treatment to evaluate continued effect of the device on local circulation in the leg.

The study will be individually controlled with each patients treated leg evaluated against the contralateral non- treated leg.

Subjective data including distance able to walk, pain and vibratory sensation threshold will also be collected and evaluated appropriately.

ELIGIBILITY:
Inclusion Criteria:

* Give appropriate written informed consent prior to participation in the study
* Have a current diagnosis of Type I or Type II Diabetes Mellitus
* Have an Ankle-Arm Index between 0.35 and 0.8 on the study limb
* Be in reasonable metabolic control, exhibited by HbA1C values of less than12% as observed by serum test results obtained within 3 months prior to the Screening Visit
* Subject and caregiver must be accessible for, and willing to comply with, the safety procedures and available for the 12 week Follow-Up Period

Exclusion Criteria:

* Clinical evidence of gangrene on any part of affected foot
* Active Charcot's foot on the study limb
* Scheduled to undergo vascular surgery, angioplasty, or thrombolysis within 30 days from the end of the study
* Malnourished as evidenced by a pre-albumin of < 11 mg/dL
* Pregnancy or lactating
* History of bleeding disorder
* Participation in another device study for the treatment of Peripheral Vascular Disease 30 days prior to Screening Visit
* Vascular procedures performed 30 days prior to Screening Visit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-10; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Chusid, PHD, Study Director — New York College of Podiatric Medicine
Locations (1):
- New York College of Podiatric Medicine, New York, New York, United States